CLINICAL TRIAL: NCT05076513
Title: A Phase 0 'Trigger' Trial of Niraparib in Newly-diagnosed Glioblastoma and Recurrent IDH1/2(+) ATRX Mutant Glioma
Brief Title: Trial of Niraparib in Participants With Newly-diagnosed Glioblastoma and Recurrent Glioma
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nader Sanai (Other)
Collaborators: Barrow Neurological Institute (Other); Ivy Brain Tumor Center (Other); University of California, San Francisco (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Nader Sanai, Chief Scientific Officer/Director, St. Joseph's Hospital and Medical Center, Phoenix
Organization: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-13
Record Dates: First submitted 2021-09-13; First posted 2021-10-13 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Glioblastoma; Glioblastoma Multiforme; Glioma; GBM; Glioma, Malignant; Glioblastoma Multiforme of Brain
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — niraparib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Presumed Newly-Diagnosed glioblastoma (Experimental): Participants undergoing resection for a presumed newly-diagnosed glioblastoma (WHO grade 4) will be treated with niraparib for 4 days prior to surgical resection. Participants who proceed to the therapeutic expansion phase of this study will receive niraparib in combination with radiation (60 Gy over 6-7 weeks, as per standard of care). Following radiotherapy, eligible study participants may receive niraparib maintenance treatment.
  Interventions: Drug: Niraparib; Radiation: Radiation therapy
- Arm B: Recurrent Glioma (Grades II-IV) (Experimental): Participants undergoing resection of a recurrent WHO Grade II, III, or IV glioma with IDH1 or IDH2 mutation and ATRX loss will be treated with niraparib for 4 days prior to a planned surgical resection. Participants who proceed to the Expansion cohort will receive niraparib in 28d cycles after surgery.
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — In Phase 0, 300mg administered orally QD for 4 days prior to resection.
  In the Expansion cohort/Maintenance phase, niraparib will be administered as described below:
  * For patients weighing <77 kg (<170 lbs) OR with a platelet count <150,000/mcL, the recommended dosage is 200 mg taken orally once daily.
  * For patients weighing ≥77 kg (≥170 lbs) AND a platelet count ≥150,000/ mcL, the recommended dosage is 300 mg taken orally once daily.
  Other Names: Zejula
Radiation: Radiation therapy — Participants in Arm A who move onto the Expansion cohort will receive 6-7 weeks of radiation therapy per standard of care.
  Arms: Arm A: Presumed Newly-Diagnosed glioblastoma

SUMMARY:
This is an open-label, multi-center Phase 0 study with an expansion phase that will enroll up to 24 participants with newly-diagnosed glioblastoma and up to 18 recurrent glioma participants with IDH mutation and ATRX loss. The trial will be composed of a Phase 0 component (subdivided into Arm A and B) and a therapeutic expansion phase. Patients with tumors demonstrating a positive PK Response (in Arm A) or a positive PD Response (in Arm B) of the Phase 0 component of the study will graduate to a therapeutic expansion phase that combines therapeutic dosing of niraparib plus standard-of-care fractionated radiotherapy (in Arm A) or niraparib monotherapy (in Arm B) until progression of disease.

ELIGIBILITY:
Inclusion Criteria:

1. Arm A participants undergoing resection for a suspected newly diagnosed glioblastoma. For Arm B, participants undergoing resection who have had a prior resection of histologically diagnosed WHO grade II-IV glioma with IDH1 or IDH2 mutation and ATRX loss.
2. Arm A participants must have measurable disease preoperatively, defined as at least 1 contrast-enhancing lesion, with 2 perpendicular measurements of at least 1 cm.
3. Ability to understand and the willingness to sign a written informed consent document (personally or by the legally authorized representative, if applicable).
4. Participant has voluntarily agreed to participate by giving written informed consent (personally or via legally authorized representative(s), and assent if applicable). Written informed consent for the protocol must be obtained prior to any screening procedures. If consent cannot be expressed in writing, it must be formally documented and witnessed, ideally via an independent trusted witness.
5. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other procedures.
6. Age ≥18 at time of consent
7. Have a performance status (PS) of ≤2 on the Eastern Cooperative Oncology (Group (ECOG) scale (Oken et al. 1982)
8. Ability to swallow oral medications.
9. Confirmed negative serum pregnancy test (β-hCG) before starting study treatment or participant who is no longer of childbearing potential due to surgical, chemical, or natural menopause. If the serum pregnancy test is completed > 7 days from Day 1, a urine pregnancy test will be done to confirm a negative result prior to Day 1 dose administration.
10. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to treatment and agreement to use such a method during study participation and for an additional 6 months after the end of treatment administration.
11. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner and for an additional 3 months after the end of treatment administration. Avoid sperm donation for duration of the study and for an additional 6 months after the end of treatment administration.
12. Agreement to adhere to Lifestyle Considerations throughout study duration.
13. Participants who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to Day 1. A washout period of at least 21 days is required between last chemotherapy and Day 1.
14. Females of child-bearing potential must agree not to breastfeed starting at screening, throughout the study period and for 6 months after final study drug administration.
15. Participant has normal blood pressure or adequately treated and controlled hypertension (Defined as systolic BP ≤140 mmHg and diastolic BP ≤90 mmHg).
16. Participant has adequate bone marrow and organ function as defined by the following laboratory values (as assessed by the local laboratory for eligibility):

    * Adequate Bone Marrow Function:

      * Absolute Neutrophil Count ≥1,500/mcL
      * Platelets (at time of surgery) ≥100,000/mcL
      * Hemoglobin ≥9.0 g/dL. Participants may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion.
    * Adequate Hepatic Function:

      * Total Bilirubin ≤1.5 X ULN. Participants with Gilbert's syndrome with a total bilirubin ≤2.0 times ULN and direct bilirubin within normal limits are permitted.
      * AST(SGOT) ≤2.5 X institutional ULN
      * ALT(SGPT) ≤2.5 X institutional ULN
    * Adequate Renal Function:

      * Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73 m2 by Chronic Disease Epidemiology Collaboration (CKD-EPI) equation
    * INR ≤1.5 x ULN

Exclusion Criteria:

1. Current use of coumarin-derived anticoagulant for treatment, prophylaxis or otherwise, that cannot be discontinued prior to surgery. Therapy with heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed.
2. Pregnancy or lactation.
3. Known allergic reactions to components of the niraparib tablet, including FD&C Yellow No. 5..
4. Active infection or fever >38.5°C requiring systemic antibiotic, antifungal or antiviral therapy within 4 weeks of Day 1.
5. Known to have active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and active and chronic hepatitis as determined by the investigator.
6. Known active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
7. Any of the following cardiovascular criteria:

   * Current evidence of cardiac ischemia
   * Current symptomatic pulmonary embolism
   * Acute myocardial infarction ≤ 6 months prior to Day 1
   * Heart failure of New York Heart Association Classification III or IV ≤ 6 months prior to Day 1 (Appendix 13.2)
   * Grade ≥ 2 ventricular arrhythmia ≤ 6 months prior to Day 1
   * Cerebral vascular accident (CVA) or transient ischemic attack (TIA) ≤ 6 months prior to Day 1
8. Participant has myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of MDS/AML.
9. Participant has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
10. Prior therapy with PARP inhibitors at a therapeutic dose.
11. Treatment with another investigational drug or other intervention within 30 days prior to enrollment or within 5 half-lives of the investigational product, whichever is longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-10-29 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Phase 0 Arm A: Total and unbound niraparib concentration in enhancing and nonenhancing tissue | Day 4 Intra-operative sample
  Tumor to plasma partition coefficients of niraparib for total (Kp) and unbound (Kp,uu) drug levels
Phase 0 Arm B: Presence of Chromosomal fusion | Day 4 Intra-operative sample
  Presence of chromosomal fusion with the cutoff CT value of 35 in niraparib treated glioma tissue with IDH and ATRX loss.
Phase 0 Expansion Arm A: Progression-free survival in participants with demonstrated PK effects | 6 months
  6 month progression-free survival (PFS6) rate measured from the time of surgery to date of recurrence.
Phase 0 Expansion Arm B: Progression-free survival in participants with demonstrated PD effects | 6 months
  6 month progression-free survival (PFS6) rate measured from the time of surgery to date of recurrence.

SECONDARY OUTCOMES:
Drug-related toxicity | 24 months
  Incidence of drug-related toxicity
Adverse events | 24 months
  Number of adverse events through study completion, assessed up to 24 months.
Deaths | 24 months
  Number and incidence of deaths
Incidence of clinical laboratory abnormalities per CTCAE | Up to 30 days after the last study dose
  Clinical laboratory abnormalities per CTCAE
Overall survival | 48 months
  Median overall survival
Phase 0 Arm A: Pharmacodynamics (PD) of niraparib | Day 4 Intra-operative Tissue
  Quantification of percentage of PAR positive cells with IHC assay or PAR concentration in tumor homogenates with an HT PARP pharmacodynamic assay II.
Phase 0 Arm B: Pharmacokinetics (PK) of niraparib | Day 4 Intra-operative Tissue
  Total and unbound niraparib concentration in Gd-enhancing and non-enhancing tumor tissue

CONTACTS AND LOCATIONS:
Overall Officials: Nader Sanai, MD, Principal Investigator — Chief Scientific Officer/Director of the Ivy Brain Tumor Center
Locations (1):
- St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ivy Brain Tumor Center Website — http://www.ivybraintumorcenter.org/